CLINICAL TRIAL: NCT05837377
Title: The Effect of Simulation-Based Training Program Designed Based on Cognitive Load Theory on Drug Administration Competency
Brief Title: Drug Administration Competency of Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14.02.2022-03/17
Record Dates: First submitted 2023-04-11; First posted 2023-05-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Nursing Student; Simulation; Cognitive Load; Competence
Keywords: cognitive load theory; Drug Administration; competency; simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control- standard medication education (Experimental): The control group will receive a traditional medication administration proficiency training program.
  Interventions: Other: Control- standard medication education
- Experiment- cognitive load theory based on medication education (Experimental): The experiment group will receive a cognitive load theory-based medication administration training program.
  Interventions: Other: Experiment- cognitive load theory based on medication education

INTERVENTIONS:
Other: Control- standard medication education — Common Procedure:
  - "Student Information and Consent Form will be obtained from the students.
  For the control group
  * Theoretical training in drug administration skills is provided.
  * Skill training: Skill training on intramuscular and subcutaneous injection and intravenous medication administration using task trainers in the simulation laboratory.
  * After the skill evaluation phase, a safe drug administration scenario will be applied.
  Arms: Control- standard medication education
Other: Experiment- cognitive load theory based on medication education — For the experiment group
  * Theoretical training will be provided based on the results of both the knowledge test and the self-efficacy test, and will be designed according to the principles of cognitive load theory.
  * Skills training: includes the necessary skill applications for students with task trainers and a virtual simulation designed according to the cognitive load theory for these skills.
  * After the skill evaluation phase, a safe drug administration scenario will be applied.
  Arms: Experiment- cognitive load theory based on medication education

SUMMARY:
The purpose of this study is to examine the effect of a simulation-based education program designed based on cognitive load theory on the development of medication administration competency of nursing students.

DETAILED DESCRIPTION:
The study was designed according to a pre-post test control group randomized controlled experimental design. During the research procedure, the medication administration competency training program will be implemented to the groups by using two different methods. In the training program will be applied to the experiment group will designed to be considered of the intrinsic, extraneous, and germane loads described in Cognitive Load Theory.

For randomization, a list of students who will be agreed to participate in the study, will be created and assigned serial numbers by a faculty other than researcher. The control and experiment groups will be formed by randomly assigning these serial numbers using a computer program (www.random.org). To prevent repeated student evaluations and potential bias, students will be tracked using their serial numbers during the data collection process.

The control group will receive the medication administration competency training program using the conventional education method.

A cognitive load theory-based medication administration competency training program will be applied to the experiment group of students. The cognitive load theory explains the amount of mental effort that is required to perform mental processes and is loaded onto memory resources. This theory helps to make learning more effective by reducing students' cognitive load, taking into account factors such as the complexity of learning materials and their presentation format. In this context, the content structuring of the training program will be determined according to the students' knowledge levels and cognitive loads that will be identified before the training program. The training program consists of theoretical education, skill training, medication administration competency virtual simulations, and scenario applications. The students' knowledge levels, cognitive loads, and medication administration competency self-assessments will be evaluated before and after the theoretical education. Skill levels will be evaluated by using structured observation tools during the skill training, and cognitive loads and clinical decision-making competency levels will be evaluated at the end of the scenario.

In data collection:

* To evaluate the knowledge levels of the control and experiment group students regarding medication administration before and after the training, the Medication Administration Knowledge Test will be used.
* To assess the psychomotor skills of students regarding medication administration, Objective Structured Clinical Examination (OSCE) checklists for medication dosage calculation and administration via intramuscular, subcutaneous, and intravenous routes will be used.
* The Medication Administration Competence Self-Assessment Form will be applied to students to assess herself on medication administration competence and its subcomponents.
* The Cognitive Load Scale will be used to determine how much mental effort the student exerts while performing tasks related to medication administration.
* The Simulation Self-Reported Cognitive Load Measurement Tool will be used to determine the cognitive, extraneous, and germane loads of the control and experiment group students after the scenario application.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old,
* Minimum 18 years old,
* To be a third or fourth-year nursing undergraduate student,
* To volunteer to participate in the research.

Exclusion Criteria:

* Inability to complete any stage of the study,
* Failure to complete data collection forms.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-11-04 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Change in medication administration knowledge level | The Medication Administration Knowledge Test will be administered before the training and again one week after the training. The change in these time intervals will be assessed.
  Medication Administration Knowledge Test scores of students in a simulation-based training programme designed according to cognitive load theory are higher than those of students in the standard training programme.
Comparison of medication administration skill performances | It will be conducted one week after the skill training. The change in these time intervals will be assessed.
  The Objective Structured Clinical Examination (OSCE) scores of students in a simulation-based training programme designed according to cognitive load theory are higher than those of students in the standard training programme.
Comparison of Clinical Decision Making Skill Level | The assessment will be conducted one week after the objective structured skill examination. The change in these time intervals will be assessed.
  Students' scores on the control list for safe drug administration scenarios in a simulation-based training programme designed according to cognitive load theory are higher than those of students in the standard training programme.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Yıldız Çelik, Phd student, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem Unıversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers BA, Franklin AE. Cognitive load experienced by nurses in simulation-based learning experiences: An integrative review. Nurse Educ Today. 2021 Apr;99:104815. doi: 10.1016/j.nedt.2021.104815. Epub 2021 Feb 20. PMID 33640776
- [Background] Fraser KL, Ayres P, Sweller J. Cognitive Load Theory for the Design of Medical Simulations. Simul Healthc. 2015 Oct;10(5):295-307. doi: 10.1097/SIH.0000000000000097. PMID 26154251
- [Background] McMullan M. Evaluation of a medication calculation mobile app using a cognitive load instructional design. Int J Med Inform. 2018 Oct;118:72-77. doi: 10.1016/j.ijmedinf.2018.07.005. Epub 2018 Jul 24. PMID 30153925
- [Background] Sweller, J. (2020). Cognitive load theory and educational technology. Educational Technology Research and Development, 68(1), 1-16. Doi: https://doi.org/10.1007/s11423-019-09701-3
- [Background] Josephsen, J. (2018). Cognitive load measurement, worked-out modeling, and simulation. Clinical Simulation in Nursing, 23, 10-15. doi:https://doi.org/10.1016/j.ecns.2018.07.004